CLINICAL TRIAL: NCT07077395
Title: Finding Links Between Hot flASHes and CardioVascular Disease
Acronym: FLASH-CV:
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Emily Lau, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025p001738
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Menopause-related Hot Flashes
Keywords: menopause; hot flashes; heart health
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- elinzanetant 120 mg daily for 12 weeks (Active Comparator)
  Interventions: Drug: elinzanetant - reference formulation
- Placebo daily for 12 weeks (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: elinzanetant - reference formulation — elinzanetant 120 mg daily x 12 weeks
  Arms: elinzanetant 120 mg daily for 12 weeks
Drug: placebo — placebo daily x 12 weeks
  Arms: Placebo daily for 12 weeks

SUMMARY:
The goal of this clinical trial is to learn if neurokinin-1/neurokinin-3 receptor antagonist elinzanetant improves blood vessel health in women with moderate to severe hot flashes. The main questions it aims to answer is does neurokinin-1/neurokinin-3 receptor antagonist elinzanetant improve blood vessel health?

ELIGIBILITY:
Inclusion Criteria:

* Age 40-65 years
* Peri- and post-menopausal women (STRAW -1 to +1)
* Moderate or high vasmotor symptom burden
* Cardiometabolic disease (as evidenced by ≥ 2 of the following):

  * Obesity (body mass index ≥ 30 kg/m2)
  * Elevated waist circumference (≥ 88 cm)
  * Elevated triglycerides (≥ 150 mg/dL or drug treatment)
  * Reduced HDL-cholesterol (<50 mg/dL or drug treatment)
  * Elevated blood pressure (≥ 130 mmHg systolic blood pressure or ≥ 85 mmHg diastolic blood pressure, or drug treatment)
  * Elevated fasting glucose (≥ 100 mg/dL or drug treatment)

Exclusion Criteria:

* Inability to provide informed consent or comply with study protocol
* Major comorbidities: cancer, end-stage renal (eGFR <45 mL/min/1.73 m2), liver or lung disease
* Concomitant use of strong or moderate cytochrome P450 3A4 inhibitors
* Elevated liver function tests (ALT, AST, and/or total bilirubin ≥2x ULN)
* Undiagnosed uterine bleeding over past 6 months

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
brachial artery flow mediated dilation | 12 weeks

SECONDARY OUTCOMES:
concentration of inflammatory protein biomarkers | 12 weeks
  * General inflammatory markers: hsCRP, IL-8, TNF-ɑ/β
  * Leukocyte adhesion markers: MCP-1, ICAM-1
  * Markers of vascular homeostasis: ANGPT1, VEGFA, HB-EGF

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lau, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol